CLINICAL TRIAL: NCT00514670
Title: A Randomized Controlled Trial of a School Disinfection and Hand Hygiene Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Study funds provided by The Clorox Company (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-01-0014
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Respiratory Infections; Gastrointestinal Diseases
Keywords: Prevention of gastrointestinal and respiratory illness
MeSH Terms: conditions — Respiratory Tract Infections; Gastrointestinal Diseases | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention classrooms received alcohol-based hand sanitizer and disinfecting wipes.
  Interventions: Other: Alcohol-based hand sanitizer & quaternary ammonium wipes
- 2 (No Intervention): No hand sanitizer or disinfecting wipes were used.

INTERVENTIONS:
Other: Alcohol-based hand sanitizer & quaternary ammonium wipes
  Arms: 1

SUMMARY:
The objective of the trial is to assess the impact of a disinfection and hand hygiene program on absenteeism in elementary school classrooms. Students in intervention classrooms will use alcohol-based hand sanitizers at school, and their classrooms will be disinfected using quaternary ammonium wipes. We hypothesize that the use of disinfectants and hand hygiene products in elementary school classrooms will reduce absenteeism.

ELIGIBILITY:
Inclusion Criteria:

* Member of a designated elementary school classroom in the Avon school system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2006-03; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Absenteeism rate due to gastrointestinal or respiratory illness during the study period. | 8 weeks

SECONDARY OUTCOMES:
Bacterial colony counts and the presence of selected viruses on classroom surfaces. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Sandora, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sandora TJ, Shih MC, Goldmann DA. Reducing absenteeism from gastrointestinal and respiratory illness in elementary school students: a randomized, controlled trial of an infection-control intervention. Pediatrics. 2008 Jun;121(6):e1555-62. doi: 10.1542/peds.2007-2597. PMID 18519460